CLINICAL TRIAL: NCT03650933
Title: A Multi-center, Randomized, Double-blind, Controlled, and Parallel Phase III Study to Compare the Efficacy and Safety of GB241 (Recombinant Anti-CD20 Human-Mouse Chimeric Monoclonal Antibody Injection, Experimental Drug) Plus CHOP Versus Rituximab Plus CHOP in Untreated Diffuse Large B-cell Lymphoma (DLBCL) Patients
Brief Title: A Study Comparing the Efficacy and Safety of G-CHOP Versus R-CHOP in Untreated Diffuse Large B-cell Lymphoma Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing Yoko Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GB241NHL3
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Diffuse Large B-Cell Lymphoma, Unspecified Site
Keywords: GB241; Rituximab; Diffuse Large B-cell Lymphoma; Non Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — R-CHOP protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-CHOP (Experimental): GB241 plus CHOP, six cycles. GB241: 375 mg/m2, IV, day 1 of each cycle; Cyclophosphamide: 750 mg/m2, IV, day 2 of each cycle; Doxorubicin: 50 mg/m2, IV, day 2 of each cycle; Vincristine: 1.4 mg/m2, up to a maximal dose of 2 mg, IV, day 2 of each cycle; Prednisone: 100 mg, po, day 2 to day 6 of each cycle.
  Interventions: Biological: G-CHOP
- R-CHOP (Active Comparator): Rituximab plus CHOP, six cycles. Rituximab: 375 mg/m2, IV, day 1 of each cycle; Cyclophosphamide: 750 mg/m2, IV, day 2 of each cycle; Doxorubicin: 50 mg/m2, IV, day 2 of each cycle; Vincristine: 1.4 mg/m2, up to a maximal dose of 2 mg, IV, day 2 of each cycle; Prednisone: 100 mg, po, day 2 to day 6 of each cycle.
  Interventions: Biological: R-CHOP

INTERVENTIONS:
Biological: G-CHOP — 6 cycles(each cycle is 3 weeks)
  Arms: G-CHOP
Biological: R-CHOP — 6 cycles(each cycle is 3 weeks)
  Arms: R-CHOP

SUMMARY:
A Multi-center, Randomized, Double-blind, Controlled, and Parallel Phase III Study to Compare the Efficacy and Safety of GB241 (Recombinant Anti-CD20 Human-Mouse Chimeric Monoclonal Antibody Injection, Experimental Drug) Plus CHOP Versus Rituximab Plus CHOP in Untreated Diffuse Large B-cell Lymphoma (DLBCL) Patients

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated CD20 Positive DLBCL.
2. International Prognostic Index (IPI) score of 0 to 2, Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
3. 18 years to 70 years; Male or female patients; Body Mass Index (BMI)≤2.13 m^2.
4. Expected survival more than 6 months.
5. At least 1 bi-dimensionally measurable lesion: Nodal lesion: Greatest transverse diameter≥1.5cm and short axis≥1.0cm; Extra-nodal lesion: Greatest transverse diameter≥1.0cm.
6. Cardiac echocardiography: LVEF≥50%.
7. Adequate hematological function: WBC≥3 x 10^9/L, HGB≥80g/L, ANC≥1.5 x 10^9/L, PLT≥75 x 10^9/L.
8. Hepatic function: TBIL≤1.5 x ULN, ALT or AST≤2.5 x ULN, ALP≤3 x ULN if with no bone marrow infiltration, Renal function: Cr≤1.5 x ULN.
9. Seronegative for HCV antibody, or HIV antibody, or hepatitis B virus surface antigen (HBsAg). HBc antibody seropositive, but HBV DNA and HBsAg negative patients may participle following consultation with a hepatitis expert regarding monitoring and use of HBV antiviral therapy, and provided they agree to receive treatment as indicated.
10. Must agree to take effective birth control methods or are not of childbearing potential. Women must agree to continue contraceptive measures within 12 months after the last treatment. Men must agree to continue contraception within 3 months after the treatment.
11. All patients must have signed an informed consent document.

Exclusion Criteria:

1. Other types of DLBCL: primary central nervous system DLBCL, primary skin DLBCL (leg type), EBV-positive DLBCL, NOS, EB virus-positive skin mucosal ulcer, chronic inflammation-related DLBCL, lymphomatoid granuloma, primary Mediastinal (thymus) large B-cell lymphoma, intravascular large B-cell lymphoma, ALK+ large B-cell lymphoma, plasmablastic lymphoma, primary exudative lymphoma, HHV8+DLBCL, NOS, Burkitt's lymph Tumor, primary testicular lymphoma。
2. Confirmed DLBCL with BCL-2 and c-MYC gene rearrangement or BCL-2, BCL-6, and c-MYC gene rearrangement by FISH. B-cell lymphomas, unclassifiable, with features intermediate between diffuse large B-cell lymphoma and Burkitt lymphoma.
3. B-cell lymphoma, unclassifiable, with features intermediate between diffuse large B-cell lymphoma and classical Hodgkin lymphoma.
4. Previous malignant tumor except cured cervical cancer,basal cell carcinoma and squamous cell skin cancer.
5. Patients who have received therapy for non-Hodgkin's lymphoma: including chemotherapy, immunotherapy; radiotherapy (excluding local radiotherapy); monoclonal antibody therapy; surgical treatment (excluding biopsy);
6. Patients who received continuous treatment of corticosteroid drugs lasting for more than 10 days. Prednisone with the dosage over 30mg/day; Other corticosteroid drugs with equal dosage.
7. Patients who received cytotoxic drugs or anti-CD20 monoclonal antibody for other diseases (such as Rheumatoid arthritis).Or received any monoclonal antibody within 3 months prior to the enrollment of the study.
8. Patients who participated in other clinical trials within 3 months prior to the enrollment of the study.
9. Patients who received attenuated or live virus vaccine within 1 month prior to the enrollment of the study.
10. Patients who received hematopoietic stimulating factors within 1 week prior to the enrollment of the study.
11. Recent major surgery within 1 month.
12. Active Infectious disease or significant infections requiring intravenous antibiotic therapy or hospitalization in the past 4 weeks (exception of tumor induced fever).
13. Known allergic reactions against human or murine monoclonal antibody, murine products, or foreign proteins.
14. Contraindicative to any drug in CHOP.
15. Patients who have significant cardiac disease, including heart disease of grade Ⅲ of Ⅳ according to the New York Heart Association(NYHA) system, or occurrence of myocardial infarction, unstable arrhythmia, unstable angina or severe hypertension in the past 6 months or peripheral nervous system(PNS) or CNS disease.
16. Suspected active tuberculosis patients.
17. Patients with serious peripheral nervous system or central nervous system disease.
18. Patients that researchers deem as not appropriate to enter the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2018-12-28 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 6 cycles(each cycle is 3 weeks)
  To evaluate the objective response rate (ORR) in patients with previously untreated Diffuse Large B-cell Lymphoma after six cycles of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China